CLINICAL TRIAL: NCT06287203
Title: Novel Prevention Intervention Program to Reduce Risky Patterns of Substance Use Among Emerging Adults
Acronym: ARFP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Danielle Dick, RWJMS, Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro2023001498; 3R01DA050721-04S1 (NIH)
Record Dates: First submitted 2024-02-21; First posted 2024-03-01 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Masking Description: Participants will not be made aware of their condition at baseline; however, they will know their condition once they receives their estimates (or not, in the case of the control condition) and are taken to their follow-up resources.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Risk estimates + Psychoeducation (Active Comparator): Participants in this condition will complete the prevention program in which individuals receive their personalized risk estimates, followed by psychoeducation about ways to reduce substance use and associated harm.
  Interventions: Behavioral: Addiction Risk Feedback Program
- Risk estimates + Online CBT Modules (Active Comparator): Participants in this condition will complete the prevention program in which individuals receive their personalized risk estimates, followed by on-line cognitive behavioral therapy (CBT)-based modules to assist with controlling substance use.
  Interventions: Behavioral: Addiction Risk Feedback Program
- Risk estimates + Genetic Counselor (Active Comparator): Participants in this condition will complete the prevention program in which individuals receive their personalized risk estimates, followed by a follow-up appointment with a genetic counselor.
  Interventions: Behavioral: Addiction Risk Feedback Program
- Waitlist Control - Psychoeducation Only (Other): Participants in this condition will not receive their personalized risk estimates until the end of the study. They will receive psychoeducation about ways to reduce substance use and associated harm at the time that the active conditions receive their estimates and associated follow-up content.
  Interventions: Behavioral: Addiction Risk Feedback Program

INTERVENTIONS:
Behavioral: Addiction Risk Feedback Program — This novel prevention/intervention program will be accessed via an on-line interactive website where individuals receive their personalized risk estimates, based on their genetic, behavioral, and environmental risk factors (part 1 of the program), accompanied by information to help them reduce risk (part 2 of the program). The information in part 2 of the program will vary between arms.

SUMMARY:
The purpose of this research study is to test whether completion of a new personalized feedback program is associated with reductions in risky substance use among emerging adults (18-25 years of age).

DETAILED DESCRIPTION:
There has been tremendous advances in gene identification. From large-scale, well-powered genome wide association studies (GWAS), polygenic scores (PGS) can now be calculated that sum risk alleles across the genome and weight them by their effect size, creating an index of genetic liability for any given individual. But genetic influences are only part of what contributes to substance use disorders; the environment also plays a critical role. Accordingly, understanding the development of substance use outcomes necessitates integrating both genetic and environmental information. The rationale for this line of research is that the integration of genetic and environmental information will provide the foundation for precision medicine, and that the provision of this personalized risk information will help prevent the development of problems and/or allow for earlier intervention before problems have become severe. Our research team is creating a new prevention/intervention program, consisting of an on-line platform for individuals to receive their personalized risk estimates for addiction risk, created by integrating information about their genetic, behavioral, and environmental risk factors followed by information about how to reduce risk.

The investigators are enrolling a sample of emerging adults (18-25 years of age) into a randomized controlled trial consisting of 4 conditions. All four conditions will involve completion of a behavioral/environmental risk survey and the provision of saliva to determine genetic risk. Three active conditions involve individuals receiving their personalized risk estimates, followed by (condition 1) psychoeducation about ways to reduce substance use and associated harm; (condition 2) the on-line CBT-based module to assist with controlling substance use; or (condition 3) a follow-up appointment with a genetic counselor (GC). The fourth condition will be a waitlist control, in which individuals will receive psychoeducation only at the time that the active conditions receive their personalized risk estimates.

At the first time point (T0), participants will be randomly selected into one of four conditions. Participants have an equal chance of being assigned to any one of the conditions. Across all conditions, the investigators will measure substance use and problems at enrollment (T0), at the time of receipt of risk estimates (~8 weeks later; or at the time other participants receive their results (~8 weeks later) in the case of control condition) (T1), 1 month (T2), and 3 months (T3) after completion of the program.

After the final survey (T3), participants in the control condition will receive their personalized risk estimates. All participants, regardless of their initial group, will be invited to receive access to the content of conditions in which they did not take part (e.g., online modules, appointment with a genetic counselor).

Findings from this study have great potential to enhance our ability to use precision medicine to prevent the development of substance use disorders and/or intervene earlier in the progression to disorder.

ELIGIBILITY:
Inclusion Criteria:

* This study is for emerging adults between 18-25 years who reside in the United States. These individuals must also be English-speaking.

Exclusion Criteria:

* Participants will be excluded from the study if they are younger than 18 years old, older than 25 years old, reside outside of the United States, or if they do not provide informed consent. These exclusion criteria have been chosen because we are targeting emerging adults (a particularly risky population in terms of substance use behaviors).

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 660 (Actual)
Dates: Start 2024-04-12 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Alcohol Consumption | 3 months
  Alcohol consumption will be measured using the Alcohol Use Disorders Identification Test (AUDIT) consumption subscale. The AUDIT-C consists of 3 items (e.g., "how often do you have a drink containing alcohol"). Items are rated on a 5-point scale. Items will be summed to create subscale totals with higher scores representing higher levels of that behavior (e.g., higher alcohol consumption. Scores can range from 0 to 12.
Alcohol Problems | 3 months
  Alcohol problems will be measured using the AUDIT problems subscale ( Bohn, Babor, & Kranzler, 1995). The AUDIT-P consists of 6 items (e.g., "how often do you have a drink containing alcohol"). Items are rated on a 5-point scale. Items will be summed to create subscale totals with higher scores representing higher levels of that behavior (e.g., higher alcohol problems). Scores can range from 0 to 24.
Drug Use Problems | 3 months
  Drug Use problems will be measured using the Drug Use Disorders Identification Test (DUDIT) scale. The DUDIT consists of 11 items (e.g., "how often do you use drugs other than alcohol"). Items are rated on a 5-point scale. Items will be summed to create subscale totals with higher scores representing higher levels of that behavior (e.g., higher drug consumption). Scores can range from 0 to 44.
Readiness to change | 3 months
  The Readiness to Change Questionnaire is a 12-item measure that provides scores for three subscales (Precontemplation, Contemplation, and Action) representing stages of change. Items (e.g., "I am trying to drink/ use other drugs less than I used to") are rated on a 5-point scale with response options ranging from "strongly disagree" to "strongly agree." Items will be summed to create three total subscale scores. Based on subscale scores, individuals will be categorized to one of the three categories. We will assess change in the percent of individuals in each category.
Future substance use intentions | 3 months
  Future substance use intentions will be assessed with three items: "how often do you plan to drink alcohol next month," "how often do you plan to get drunk next month," and "how often do you plan to use drugs next month" with response options of "less than last month," "the same as last month," and "more than last month." We will assess change in the percent of individuals in each category (less, same, more than last month) for all three items.

SECONDARY OUTCOMES:
Worry About Substance Use Disorders | Baseline to 3 months
  An adapted version of the Cancer Worry Scale will be used to assess worry about developing substance use disorders within the past 30-days. The scale consists of 8 items (e.g., "How often do you worry about developing alcohol or other drug use disorder?") rated on a 4-point scale. Items will be summed to create a total scale score with higher scores reflecting higher levels of worry about substance use disorders.
Perceived Susceptibility | 3 months
  Perceived susceptibility of developing alcohol use or other drug use disorder will be assessed using the Health Beliefs about Mental Illness Instrument (Saleeby, 2000). The scale consists of 5-items (e.g., "my chances of having alcohol or other drug problems are great") rated on a 5-point scale with response options ranging from "strongly agree" to "strongly disagree." Items will be summed to create a total scale score with higher scores reflecting higher perceived susceptibility for substance use disorders.
Well-Being | 3 months
  Well-being will be assessed with the Mental Health Continuum-Short Form. The scale consists of 14-items which assess aspects of positive mental health (e.g., "I felt happy") over the past 30-days. The items are rated on a 6-point scale with response options ranging from "never" to "every day." Items will be summed to create a total scale score with higher scores reflecting higher levels of positive well-being
Anxiety and Depressive Symptoms | Baseline to 3 months
  Abbreviated scales from the Symptom Checklist-90 will be used to assess anxiety and depressive symptoms occurring within the past 30-days. The anxiety (e.g., "nervousness or shakiness inside") and depressive symptoms (e.g., "feeling no interest in things) subscales consist of four items each. Items are rated on a 5-point Likert-type scale with response options ranging from "not at all to "extremely." Items will be summed to create total subscale scores with higher scores reflecting higher levels of anxiety and depressive symptoms.
Addiction Risk Program Satisfaction | immediately after the intervention
  Satisfaction with the addiction risk program will be assessed with 12 items after participants receive their personalized risk estimates. Example items include "I learned new information as part of this program," "I enjoyed receiving my personalized risk profile," and "The online delivery method of the information was convenient." The items are rated on a 5-point scale with response options ranging from "strongly agree" to "strongly disagree."This will only be administered to the three active interventions.
Feelings About Results | immediately after the intervention
  Feelings about receiving results will be assessed with an adapted version of the Feelings About Genomic Testing Results Questionnaire. 10 items will be used to measure how participants feel about their personalized risk estimates. The items will be rated on a 5-point scale with response options ranging from "not at all" to "a great deal." Items will be summed to create a total scale score, with higher scores reflecting more positive feelings about receiving genetic test results. This will only be administered to the three active interventions.
Satisfaction with the Assigned Conditions | 3 months
  Satisfaction with the three conditions (psychoeducation, CBT, and genetic counseling) will be assessed with 10 items. Beyond the name of the condition referred to in each of the items ("education content," "modules," and "genetic counseling", respectively) the satisfaction items are the same for each of the three conditions (e.g., "I learned useful information as part of the modules"). The items are rated on a 5-point scale with response options ranging from "strongly agree" to "strongly disagree." The satisfaction items will be administered to the waitlist control in the T1part 2 survey, and it will be administered to the three active conditions in the T2 and T3 follow-up surveys. If the participant completed the satisfaction items at T2, they will not receive them again at T3.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Dick, PhD, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- Rutgers Robert Wood Johnson Medical School, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Bohn MJ, Babor TF, Kranzler HR. The Alcohol Use Disorders Identification Test (AUDIT): validation of a screening instrument for use in medical settings. J Stud Alcohol. 1995 Jul;56(4):423-32. doi: 10.15288/jsa.1995.56.423. PMID 7674678
- [Background] Berman AH, Bergman H, Palmstierna T, Schlyter F. Evaluation of the Drug Use Disorders Identification Test (DUDIT) in criminal justice and detoxification settings and in a Swedish population sample. Eur Addict Res. 2005;11(1):22-31. doi: 10.1159/000081413. PMID 15608468
- [Background] Dar-Nimrod I, Zuckerman M, Duberstein PR. The effects of learning about one's own genetic susceptibility to alcoholism: a randomized experiment. Genet Med. 2013 Feb;15(2):132-8. doi: 10.1038/gim.2012.111. Epub 2012 Aug 30. PMID 22935722
- [Background] Derogatis LR, Lipman RS, Covi L. SCL-90: an outpatient psychiatric rating scale--preliminary report. Psychopharmacol Bull. 1973 Jan;9(1):13-28. No abstract available. PMID 4682398
- [Background] Keyes CLM. Brief description of the mental health continuum short form (MHC-SF). 2009. http://www.sociology.emory.edu/ckeyes/
- [Background] Heather N, Rollnick S, Bell A. Predictive validity of the Readiness to Change Questionnaire. Addiction. 1993 Dec;88(12):1667-77. doi: 10.1111/j.1360-0443.1993.tb02042.x. PMID 8130706
- [Background] Custers JA, van den Berg SW, van Laarhoven HW, Bleiker EM, Gielissen MF, Prins JB. The Cancer Worry Scale: detecting fear of recurrence in breast cancer survivors. Cancer Nurs. 2014 Jan-Feb;37(1):E44-50. doi: 10.1097/NCC.0b013e3182813a17. PMID 23448956
- [Background] Saleeby JR. Health beliefs about mental illness: An instrument development study. American Journal of Health Behavior. 2000;24(2):83-95.
- [Background] Li M, Bennette CS, Amendola LM, Ragan Hart M, Heagerty P, Comstock B, Tarczy-Hornoch P, Fullerton SM, Regier DA, Burke W, Trinidad SB, Jarvik GP, Veenstra DL, Patrick DL. The Feelings About genomiC Testing Results (FACToR) Questionnaire: Development and Preliminary Validation. J Genet Couns. 2019 Apr;28(2):477-490. doi: 10.1007/s10897-018-0286-9. Epub 2018 Dec 14. PMID 30964586

DOCUMENTS (1):
  • Informed Consent Form (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/03/NCT06287203/ICF_000.pdf